CLINICAL TRIAL: NCT05134259
Title: The Role of Repetitive Transcranial Magnetic Stimulation in Spastic Hemiplegic Cerebral Palsy in a Sample of Egyptian Children
Brief Title: rTMS in Spastic Hemiplegic Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Fattah Muhammad, physician, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000043
Record Dates: First submitted 2021-11-20; First posted 2021-11-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The children in this group will receive traditional treatment of hemiplegic CP including medical treatment and physiotherapy in addition to repetitive transcranial magnetic stimulation sessions for 4 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Control Group (No Intervention): The children in this group will receive traditional treatment of hemiplegic CP including medical treatment and physiotherapy for 4 weeks.

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — TMS device will deliver repetitive trains of magnetic pulses using Magstim Rapid 2 with angulated figure of eight shaped coil. The device comprised two-channel Neuro-EMG-MS digital system for determining the motor threshold of the patients that will be used for establishing the threshold intensity for stimulation. The figure of eight-shaped coil generated a magnetic field of up to 4 Tesla that penetrates the cranium, enters into the soft tissue of the brain and henceforth stimulates the motor neurons.
  Arms: Study Group

SUMMARY:
The aim of the work is to study the role of repetitive transcranial magnetic stimulation (rTMS) in spastic hemiplegic cerebral palsy in a Sample of Egyptian Children.

DETAILED DESCRIPTION:
Prior to start of rTMS therapy, Gross Motor Function Classification System (GMFCS) will be employed on the participants to classify gross motor function. Also, Modified Ashworth Scale (MAS) scoring will be employed on the participants to access spasticity on selected muscles namely, hamstring, soleus, gastrocnemius and adductor of lower limb; and bicep, supinator and wrist extensor of upper limb.

rTMS frequency of 10 Hz will be delivered to each of the participants in the study group for 15 minutes per session. Each session will be administered once daily for 2 days a week for 4 weeks. 1500 pulses (50 pulses per train with total 30 trains having inter- train delay of 25 seconds) per session will be provided with the coil placed on the contralateral primary motor cortex (M1) which is known to produce modulatory effect on muscle tightness of the limbs (Rajak et al. 2017). rTMS frequency of 10 Hz was kept constant based on previous studies with 5 Hz and 10 Hz (Anttila et al. 2008) (Rossi 2009).

Each session will be followed by physical therapy (PT) according to physiotherapy protocol. After completion of therapeutic programs (after 4 weeks), the participants will be asked to undergo post assessment of Gross Motor Function Classification System (GMFCS), and Modified Ashworth Scale (MAS) scoring on exactly the same muscles as recorded previously. Both PT and rTMS sessions will be administered by trained professionals who was kept blinded to the research protocols used in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate.
2. Age group between 4 and 18 years.
3. They are able to walk with limitation or holding on according to Gross Motor Function classification System (GMFCS) (level II, III, IV).
4. All patients have mild to moderate spasticity according to modified Ashworth scale (Grade 1, 1+,2).

Exclusion Criteria:

* All Children with:

  1. Perceptual defects (IQ<70).
  2. Use of botulinum toxin in the past 4 months.
  3. Convulsions.
  4. Other peripheral or central nervous system dysfunction.
  5. Fixed deformities in lower limbs.
  6. Clinically suspected active inflammatory or pathologic changes in lower limb joints during the previous 6 months.
  7. Clinically suspected active medical problems, such as pneumonia, meningitis, encephalitis, upper gastrointestinal bleeding, or urinary tract infection.
  8. Metabolic disorders, such as inborn error of metabolism, electrolyte, and endocrine disorders.
  9. Metallic implants.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in muscle spasticity | 1 week following end of treatment
  Assessment tools: Modified Ashworth Scale. It grades muscle spasticity between 0 to 4. Higher score mean a worse outcome.

SECONDARY OUTCOMES:
Change in gross motor function | 1 week following end of treatment
  Gross Motor Function Classification System (GMFCS). It includes five levels and four age bands. Classifications are made based on the child's self-initiated movements with emphasis on sitting and walking. Higher score mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M. Emam, professor, Study Chair — Faculty of Medicine, Al-Azhar University
Locations (1):
- Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akpinar P. Vitamin D status of children with cerebral palsy: Should vitamin D levels be checked in children with cerebral palsy? North Clin Istanb. 2018 Aug 8;5(4):341-347. doi: 10.14744/nci.2017.09581. PMID 30860516
- [Background] Allen CH, Kluger BM, Buard I. Safety of Transcranial Magnetic Stimulation in Children: A Systematic Review of the Literature. Pediatr Neurol. 2017 Mar;68:3-17. doi: 10.1016/j.pediatrneurol.2016.12.009. Epub 2017 Jan 4. PMID 28216033
- [Background] Anttila H, Autti-Ramo I, Suoranta J, Makela M, Malmivaara A. Effectiveness of physical therapy interventions for children with cerebral palsy: a systematic review. BMC Pediatr. 2008 Apr 24;8:14. doi: 10.1186/1471-2431-8-14. PMID 18435840
- [Background] Gray L, Ng H, Bartlett D. The gross motor function classification system: an update on impact and clinical utility. Pediatr Phys Ther. 2010 Fall;22(3):315-20. doi: 10.1097/PEP.0b013e3181ea8e52. PMID 20699783
- [Background] Gunduz A, Kumru H, Pascual-Leone A. Outcomes in spasticity after repetitive transcranial magnetic and transcranial direct current stimulations. Neural Regen Res. 2014 Apr 1;9(7):712-8. doi: 10.4103/1673-5374.131574. PMID 25206878
- [Background] Korzeniewski SJ, Slaughter J, Lenski M, Haak P, Paneth N. The complex aetiology of cerebral palsy. Nat Rev Neurol. 2018 Sep;14(9):528-543. doi: 10.1038/s41582-018-0043-6. PMID 30104744
- [Background] Laakso I, Murakami T, Hirata A, Ugawa Y. Where and what TMS activates: Experiments and modeling. Brain Stimul. 2018 Jan-Feb;11(1):166-174. doi: 10.1016/j.brs.2017.09.011. Epub 2017 Sep 27. PMID 29030110
- [Background] Michael-Asalu A, Taylor G, Campbell H, Lelea LL, Kirby RS. Cerebral Palsy: Diagnosis, Epidemiology, Genetics, and Clinical Update. Adv Pediatr. 2019 Aug;66:189-208. doi: 10.1016/j.yapd.2019.04.002. Epub 2019 May 15. No abstract available. PMID 31230694
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Background] Patel DR, Neelakantan M, Pandher K, Merrick J. Cerebral palsy in children: a clinical overview. Transl Pediatr. 2020 Feb;9(Suppl 1):S125-S135. doi: 10.21037/tp.2020.01.01. PMID 32206590
- [Background] Rajak BL, Gupta M, Bhatia D, Mukherjee A. Increasing Number of Therapy Sessions of Repetitive Transcranial Magnetic Stimulation Improves Motor Development by Reducing Muscle Spasticity in Cerebral Palsy Children. Ann Indian Acad Neurol. 2019 Jul-Sep;22(3):302-307. doi: 10.4103/aian.AIAN_102_18. PMID 31359942
- [Background] Gupta M, Rajak BL, Bhatia D, Mukherjee A. Neuromodulatory effect of repetitive transcranial magnetic stimulation pulses on functional motor performances of spastic cerebral palsy children. J Med Eng Technol. 2018 Jul;42(5):352-358. doi: 10.1080/03091902.2018.1510555. Epub 2018 Sep 3. PMID 30175934
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552